CLINICAL TRIAL: NCT05452161
Title: Effects of Interdisciplinary Preoperative Preparation, Education, and Follow-up Sessions on Length of Stay in Hospital and Clinical Outcomes of Patients Undergoing Total Hip or Knee Replacement Surgery.
Brief Title: Effects of Preoperative Education, and Follow-up Sessions of Patients With Total Hip and Knee Arthroplasty (ESIPPES)
Acronym: ESIPPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haute Ecole de Santé Vaud (Other)
Responsible Party: Principal Investigator, Claude Pichonnaz, Associate Professor UAS, Ph.D., Haute Ecole de Santé Vaud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESIPPES
Record Dates: First submitted 2022-06-27; First posted 2022-07-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: knee; hip; replacement; arthroplasty; patient education; preoperative care; perioperative care; interdisciplinary intervention; physiotherapy; nursing
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled trial, comparing 3 modes of intervention. A single-center study conducted at the Musculoskeletal Department of the University of Lausanne The control group receives the standard care in place in the department, including only a group information session (1/3 of the sample).
  Intervention group A receives, in addition to a group information session, an individualized preparation and education session (2/3 of the sample).
  Intervention group B receives, in addition to a group information session, an individualized preparation and education session, and a remote postoperative follow-up (1/2 of group A = 1/3 of the sample).
  Patients are randomly assigned to their group based on their order of arrival. Hip and knee surgery patients are randomized separately, to keep the same proportions in each of the three groups. Block randomisation will be carried out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care (Active Comparator): Control group receives the standard care in place in the service, a group information session about knee/hip arthroplasty surgery.
  Interventions: Other: Control group
- Standard care + individualized patient-centered preparation and education session (Experimental): Intervention group A receives, in addition to standard care, an individualized patient-centered preparation and education session
  Interventions: Other: Intervention group A
- Standard care + individualized patient-centered preparation and education session + remote follow-up (Experimental): Intervention group B receives, in addition to standard care and an individualized patient-centered preparation and education session, a remote postoperative follow-up
  Interventions: Other: Intervention group B

INTERVENTIONS:
Other: Control group — All patients follow only the standard care of the department, which includes a preoperative group session of 1h30, with 15 to 30 participants, 6 to 8 weeks before the operation The objectives of these sessions are to inform the patients in a general way about the operation, its preparation and the postoperative process in order to standardize the information received. The content includes general information from the surgeon, explanations related to the course and management of patients by the various professionals (nurse, surgeon, anesthesist, physiotherapist, ergotherapist and liaison-nurse).
  Arms: Standard care
Other: Intervention group A — The day of the preparatory surgical consultation (CPC), the patient has a 30 minute patient-centered education session by a physiotherapist and a 30 minute patient-centered education session by a nurse. The physiotherapist's session addresses the technical skills to be mastered postoperatively (crutching, stairs, exercises), the course of postoperative rehabilitation, the patient's role in the rehabilitation process, the questions still remaining on this subject and the patient's perspective concerning the rehabilitation (degree and sources of anxiety, expectations of follow-up and results, degree of self-efficacy). The nursing intervention addresses the postoperative pain management, the patient's role in pain management, the care pathway, the organization of the return home and the postoperative follow-up.
  Arms: Standard care + individualized patient-centered preparation and education session
Other: Intervention group B — In addition to intervention A, patients receive a interdisciplinary intervention of three 10-15 minute phone or video conferences between the patient, a physiotherapist and a nurse.
  The aim of these interviews is to identify the patient's difficulties in the living environment, to detect possible postoperative complications and to provide advice on practical aspects (e.g. ability to perform activities), therapeutic aspects (e.g. exercises to be performed, medication), pain management, interpretation of symptoms and subjective needs (e.g. need for support). Advice on rehabilitation and care is individualized according to the results of the questionnaires administered on the day of the pre-surgical consultation and those administered at discharge, as well as the needs of the moment discussed with the patient. Any suspected complication is reported to the operating physician for appropriate management.
  Arms: Standard care + individualized patient-centered preparation and education session + remote follow-up

SUMMARY:
The shortening of the length of stay implies rethinking the perioperative management (around the operative period), which precedes and immediately follows the operation, in order to ensure a good preparation of the patient and an adequate postoperative follow-up.

The aim of this study is to evaluate the effect on the length of stay of adding an individualized preoperative preparation and education session to the current protocol in the musculoskeletal department at the CHUV in patients undergoing total hip or knee replacement surgery.

The implementation of a targeted, low-impact immediate postoperative follow-up could contribute to improving the detection of complications, preventing avoidable readmissions, improving the management of pain and adverse events, supporting the patient and responding to difficulties encountered in the patient's living environment. However, the actual added value for the patient and for the healthcare system has yet to be specified. As patients' needs and resources vary, it would also be useful to better determine the profile of patients for whom a pre- and postoperative session provides significant added value.

DETAILED DESCRIPTION:
In Switzerland, in 2017,12.4% of the Swiss population suffered from osteoarthritis. In 2019, the SIRIS hip and knee implant registry recorded 20,077 total hip replacement (THR) and 15,453 total knee replacement (TKR) implants in Switzerland.

The placement of THR and TKR is one of the major activities of the Department of the Musculoskeletal System of the CHUV (DAL-CHUV), with respectively 282 THR and 218 TKR placed in 2019.

The improvement of global practices in prosthetic surgery, the pressure on health costs and the shift to ambulatory care have led to a shortening of the length of stay.

The shortening of the length of stay implies rethinking the perioperative care (around the operative period), which precedes and immediately follows the operation, in order to ensure good preparation of the patient and adequate postoperative follow-up.

Currently, patients of the DAL-CHUV participate in a pre-operative information session (only before the operation) in a group that informs patients about the procedure, its preparation and its implications in general.

Pre-operative management is described in the literature as a multidisciplinary approach to cover all aspects to be taken into consideration in the patient, and thus prepare him/her in an optimal way for the operation and the recovery phase that will follow. Pre-operative or peri-operative rehabilitation is a broader concept of optimized recovery, which involves addressing the entire peri-operative process. Thus, the patient's health status, nutritional status, the operative and immediate postoperative process, pain management, prevention of complications and definition of relevant criteria for return home are all elements to be taken into account in an interdisciplinary manner to optimize the entire perioperative process.

The main objective of the study is to evaluate in patients undergoing total hip (THR) or knee (TKR) replacement surgery whether the addition of an individualized pre- and peri-operative preparation and education session to the existing protocol in the DAL-CHUV, provided by physiotherapists and nursing staff, has an effect on length of stay, hospital indicators, and objective and subjective clinical indicators.

The main hypothesis is that targeted pre- and peri-operative information adapted to the needs of patients would contribute to a decrease in length of stay.

The secondary indicators are readmission rate, discharge destination, postoperative pain, complications, joint function and mobility, anxiety and depression, pain representation, expectations of the prosthesis, satisfaction with care and quality of life. The hypothesis is that these indicators will be improved by the intervention.

The 1st secondary objective of the study is to evaluate in patients operated on for a total hip or knee prosthesis who have benefited from the preparation and education session whether the addition of a remote postoperative follow-up (3 telephone interviews or videoconferences during the 1st postoperative week after discharge) has additional effects on the measured indicators. The hypothesis is that the intervention will provide an additional beneficial effect for these indicators.

The 2nd secondary objective is to identify whether the effect of the pre- and postoperative interventions differs according to the characteristics of the population and the operation (THR or TKR). This secondary analysis will help to better identify the categories of populations for which the proposed peri-operative interventions are useful. The hypothesis is that the effects are dependent on patient characteristics, such as age, education level, or comorbidities for example.

Recruitment was carried out within the DAL-CHUV, based on consultation of the list of patients scheduled for a primary THR or TKR operation, and then consultation of their medical records by the study's scientific collaborator, who is also a collaborating physiotherapist at the CHUV, to verify the inclusion and exclusion criteria.

At the pre-operative information session (PIS), the important points of the study are presented orally and the consent forms of the patients who have made their decision are collected. An individual discussion will take place with those who wish to have more information about the study. The consent form is kept as part of the study files.

Those who wish to have time to reflect after the PIS will be contacted again the following week to find out their decision. They will hand in their approved consent form at the time of the pre-surgical consultation (PSC).

Once their decision is known, patients will be assigned to their group according to the randomization list.

The information of the intervention group A and B (preop and postop) does not imply any additional travel for the patient, there is only additional time dedicated to them during the PSC for the preop (group A and B) and postop (group B). The time for filling in the forms is essentially included in the consultation time (waiting time for the PSC and 6th week control), the hospital stay (day of discharge), as well as at home (2 weeks post-operatively).

The duration of the study per participant is approximately 10 weeks, PSC intervention approximately 3 weeks before the intervention, last follow-up 6 weeks after the intervention during the routine follow-up consultation at DAL-CHUV.

Descriptive statistics will be carried out for all quantitative variables of the study (means and standard deviation or medians and interquartile ranges, frequency, depending on the continuous, ordinal or nominal nature of the data), as well as graphical representations (box plot, histograms, pie chart).

The qualitative data collected will be grouped by theme and their frequency of occurrence will be analyzed (e.g. nature and frequency of occurrence of difficulties at home) For the main analysis, a Student's t test comparing the length of hospitalization between control and intervention groups will be applied. Linear regression models will then be used to adjust the difference between the groups for various potentially confounding factors (e.g. age, comorbidities, etc.). A sample size of N=200 allows for many adjustments to be included, with up to 13 parameters being estimated using the 15 observations per parameter rule.

To assess group differences in post-hospitalization measured values, linear mixed models will be used. This allows for repeated measurements (3 measurements per patient) while adjusting for various confounding factors.

A stratified analysis will be performed to differentiate the effects of the interventions in the various subpopulations of interest (e.g. age, comorbidities...), in order to identify those who particularly benefit from the tested interventions.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients admitted to the CHUV musculoskeletal department during the study period
* primary total hip replacement or primary total knee replacement
* a Risk Assessment and Prediction Tool (RAPT) score >6

Exclusion Criteria:

* a RAPT score <6,
* knee/hip arthroplasty revision surgery
* inability to give informed consent or answer questionnaires knowledgeably due to language or cognitive impairment as reported in the medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Hospital stay | 2 weeks post-surgery
  Length of hospital stay (days)

SECONDARY OUTCOMES:
Readmission rate | Consultation 6 weeks post-op
  frequency of readmission in percent
Destination at discharge | 2 weeks post-surgery
  home, rehabilitation center, nursing home for the elderly, other hospital
Postoperative pain | Day of pre-operative surgical consultation, 3 days post-surgery, Control at 2 weeks post-surgery, Medical consultation at 6 weeks post-surgery
  numerical pain scale, minimum score = 0, maximum score = 10, higher score is worse
Complications | 3 days post-surgery, Control at 2 weeks post-surgery, Medical consultation 6 weeks post-surgery
  complication type (thrombosis, pneumonia, infection, others) and rate (percent)
Joint function of hip or knee | Day of pre-operative surgical consultation, Control at 2 weeks post-surgery, Medical consultation 6 weeks post-surgery
  Western Ontario and McMaster University Osteoarthritis Index (WOMAC) (knee and hip), minimum score = 0, maximum score = 96, higher score is worse
Joint function of hip | Day of pre-operative surgical consultation, Control at 2 weeks post-surgery, Medical consultation 6 weeks post-surgery
  Hip disability and Osteoarthritis Outcome Score (HOOS-JR), minimum score = 0, maximum score = 100, higher score is worse
Joint function of knee | Day of pre-operative surgical consultation, Control at 2 weeks post-surgery, Medical consultation 6 weeks post-surgery
  Knee injury and Osteoarthritis Outcome (KOOS-JR), minimum score = 0, maximum score = 100, higher score is worse
Mobility of hip or knee | Day of pre-operative surgical consultation, Control at 2 weeks post-surgery, Medical consultation 6 weeks post-surgery
  Mobility by the degrees of the joint, min score = 0, maximum score = 360, higher score is better
Anxiety and Depression | Day of pre-operative surgical consultation, 3 days post-surgery, Control at 2 weeks post-surgery, Medical consultation 6 weeks post-surgery
  Hospital Anxiety and Depression scale (HAD), minimum score = 0, maximum score = 21 for anxiety and 21 for depression, higher score is worse
Representation of pain | Day of pre-operative surgical consultation, Control at 2 weeks post-surgery, Medical consultation 6 weeks post-surgery
  Pain Catastrophizing Scale (PCS), minimum score = 0, maximum score = 52, higher score is worse
Expectations concerning the prosthesis and subjective function | Day of pre-operative surgical consultation, 3 days post-surgery
  Hospital for Special Surgery (HSS) Hip/Knee Replacement Expectations Questionnaires, minimum score = 0, maximum score = 76, higher score means higher expectations
Satisfaction with care | Control at 2 weeks post-surgery
  Questionnaire from the Swiss National Association for Quality Development in Hospitals and Clinics (ANQ), minimum score = 0, maximum score = 5, higher score is worse, no total score, each question is analysed separately
Quality of life EuroQol 5 Dimensions (EQ-5D) questionnaire | Day of pre-operative surgical consultation and Consultation 6 weeks post-op
  Subjective indicators: questionnaire of quality of life EQ-5D, minimum score = 0, maximum score = 100, higher score is better

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichonnaz, Principal Investigator — Haute Ecole de Santé Vaud
Locations (1):
- University Hospital of Lausanne CHUV - UNIL, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weyker PD, Webb CA. Establishing a patient centered, outpatient total joint home recovery program within an integrated healthcare system. Pain Manag. 2020 Jan;10(1):23-41. doi: 10.2217/pmt-2019-0040. Epub 2019 Dec 19. PMID 31852383
- [Background] Feng JE, Novikov D, Anoushiravani AA, Schwarzkopf R. Total knee arthroplasty: improving outcomes with a multidisciplinary approach. J Multidiscip Healthc. 2018 Jan 25;11:63-73. doi: 10.2147/JMDH.S140550. eCollection 2018. PMID 29416347
- [Background] Wainwright TW, Gill M, McDonald DA, Middleton RG, Reed M, Sahota O, Yates P, Ljungqvist O. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Feb;91(1):3-19. doi: 10.1080/17453674.2019.1683790. Epub 2019 Oct 30. PMID 31663402
- [Background] Carli F, Scheede-Bergdahl C. Prehabilitation to enhance perioperative care. Anesthesiol Clin. 2015 Mar;33(1):17-33. doi: 10.1016/j.anclin.2014.11.002. Epub 2015 Jan 9. PMID 25701926
- See also: SIRIS Swiss National Joint Registry, Hip and Knee 2021 — https://www.siris-implant.ch/fr/Downloads&category=16